CLINICAL TRIAL: NCT01683682
Title: An Open Label Phase I Dose Escalation Trial of Oral BIBF 1120 in Combination With Intravenous Carboplatin and Vinorelbine in Elderly Patients With Advanced Non-Small Cell Lung Cancer - Stage IV
Brief Title: An Dose Escalation Trial of Oral BIBF 1120 in Combination With Intravenous Carboplatin and Vinorelbine in Elderly Patients With Advanced Non-Small Cell Lung Cancer - Stage IV (VENUS-2)
Acronym: VENUS-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aktion Bronchialkarzinom e.V. (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABC-2011-NSCLC-04; 2011-002141-36 (EudraCT Number)
Record Dates: First submitted 2012-08-28; First posted 2012-09-12 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small Lung Cancer; NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — nintedanib; Vinorelbine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BIBF 1120, Vinorelbine, Carboplatin (Experimental): To determine the 'Maximum Toleraetd Dose', dose escalation for BIBF 1120 will be conducted following the 3 + 3 design. A cohort of three patients will be treated at the starting dose level 150mg bid and observed until the end of the first cycle.
  Under certain conditions the dose level will be escalated to 200mg bid in a second cohort.
  Interventions: Drug: BIBF 1120; Drug: Vinorelbine; Drug: Carboplatin

INTERVENTIONS:
Drug: BIBF 1120 — 2 x 150 mg capsules, oral, daily (Start dose)
Drug: Vinorelbine — 25 mg/m2 i.v. on day 1 and 8 (three-week cycle)
Drug: Carboplatin — AUC 5 i.v. on day 1 (three-week cycle)

SUMMARY:
To investigate the maximum tolerated dose of BIBF 1120 and safety in escalating doses administered with Vinorelbine i.v. and Carboplatin i.v. in elderly patients with advanced Non-Small Lung Cancer (Stage IV).

DETAILED DESCRIPTION:
Patients older than 70 years could be enrolled in this clinical trial. The trial is being carried out in two trial centres in Germany.

For the planned sample size it is assumed that two different dosage groups are needed with 6 patients on each dosage group with the option to deescalate the first dosage. Altogether this leads to an estimated sample size of maximal 18 patients.

* Duration of treatment/patient: up to 6 month
* Follow Up: at least 6 month

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed Non-Small-Cell lung cancer (NSCLC)
* Tumor stage IV (UICC 7th Version)
* ECOG <2
* Age > 70 years
* No previous chemotherapy for stage IV NSCLC (UICC 7th Version)
* Adjuvant or neoadjuvant chemotherapy for NSCLC must be completed at least one year prior to study enrolment (from end of chemotherapy)
* Patients with prior radiation therapy may be eligible for this study if they meet the following guidelines:

  * Previous radiation therapy is allowed to <25% of the bone marrow (Cristy and Eckerman 1987), but should have been limited and must not have included whole pelvis radiation.
  * Patients must have recovered from the toxic effects of the treatment prior to study enrolment (except for alopecia).
  * Prior thoracic radiotherapy must be completed 30 days before study enrolment.
  * Lesions that have been irradiated cannot be included as sites of measurable disease unless clear tumour progression has been documented in these lesions since the end of radiation therapy.
  * Palliative extrathoracic radiotherapy to pre-existing lesions may continue on study; however, these lesions may not be included as sites of measurable disease.
* Adequate haematological laboratory parameters:

  * Haemoglobin ≥9 g/dl
  * WBC ≥3.000/µl
  * Platelets ≥ 100.000/µl
  * Neutrophil count > 1,500/µl
* Adequate renal laboratory parameters

  * Creatinine ≤1,9 mg/dl
  * Creatinine Clearance > 45 ml/min
* Adequate hepatic function

  * Total bilirubin within normal range
  * Total bilirubin < 1.5 x ULN (patients with liver metastasis)
  * ALT < 1.5 x ULN
  * ALT < 2.5 x ULN (patients with liver metastasis)
  * AST < 1.5 x ULN
  * AST < 2.5 x ULN (patients with liver metastasis)
  * Alk. phosphatase < 3 x ULN
  * LDH < 5 x ULN ULN = Upper Limit Of Normal (ULN)
* Other lab parameters:

  * Proteinuria < CTCAE grade 2
  * Prothrombin time and/or partial thromboplastin time < 50 % deviation from normal limits
* Informed consent, personally signed and dated to participate in the study
* Male patients enrolled in this trial must use adequate barrier birth control measures during the course of treatment and for at least 3 months after the last administration of study therapy
* Life expectancy at least 3 months

Exclusion Criteria:

* Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which could jeopardise compliance with the protocol
* Serious infections requiring systemic antibiotic (e.g antiviral, antimicrobial, antifungal) therapy
* Serious, non-healing wound, ulcer or bone fracture or major injuries and/or surgery within 4 weeks of trial inclusion, or planned surgical procedures during the trial period.
* Investigational drug therapy outside of this trial during or within 4 weeks of study entry
* Known hypersensitivity to the trial drugs or their excipients.
* History of other malignancies in the last 5 years, in particular those which could affect compliance with the protocol or interpretation of results. Patients with adequately treated basal or squamous cell skin cancer are generally eligible.
* Serious concomitant disease, especially those that would limit compliance with trial requirements or which are considered relevant for the evaluation of the efficacy or safety of the trial drug, such as neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with trial participation or trial drug administration, and in the judgment of the investigator would make the patient inappropriate for entry into the trial.
* Significant cardiovascular diseases (i.e. uncontrolled hypertension, unstable angina, history of infarction within past 9 months, congestive heart failure >NYHA II)
* Known inherited predisposition to bleeds or to thrombosis.
* Patient with brain metastases that are symptomatic and/or require therapy.
* Therapeutic anticoagulation (except low dose heparin and/or heparin flush as needed for maintenance of an indwelling intravenous device) or antiplatelet therapy (except for chronic low-dose therapy with acetylsalicylic acid ≤ 325mg per day)
* History of major thrombotic events or clinically relevant major bleeding event in the past 6 months (excluding central venous catheter thrombosis and peripheral deep vein thrombosis below the joint space of the knee)
* Current peripheral neuropathy ≥ CTCAE grade 2 except due to trauma
* Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug
* Active alcohol or drug abuse.
* Men who are sexually active and unwilling to use a medically acceptable method of contraception
* Leptomeningeal disease
* Radiographic evidence of cavitary or necrotic tumours
* Centrally located tumours with radiographic evidence (CT or MRI) of local invasion of major blood vessels

Min Age: 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To investigate the maximum tolerated dose of BIBF 1120 | Cycle 1 day 1, day 8, day 15; Cycle 2 day 1, day 8, day 15; Cycle 3 day 1, day 8, day 15; Cycle 4 day 1, day 8, day 15; day 84

SECONDARY OUTCOMES:
Incidence of adverse events | Cycle 1 day 1, day 8, day 15; Cycle 2 day 1, day 8, day 15; Cycle 3 day 1, day 8, day 15; Cycle 4 day 1, day 8, day 15; day 84
Response Rate | Day 43 (prior start of cycle 3), day 84

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Martin Wolf, MD, Principal Investigator — Klinikum Kassel GmbH, D-34125 Kassel; Prof. Dr. Rudolf M. Huber, MD, Study Chair — Klinikum der Universität München, D-80336 München
Locations (2):
- Germany (2):
  - Krankenhaus Großhansdorf, Großhansdorf
  - Klinikum Kassel GmbH, Kassel